CLINICAL TRIAL: NCT05790538
Title: PATTERN: Predicting the Impact of Treatment Toxicities on Health During Cancer
Brief Title: Predicting the Impact of Treatment Toxicities on Health During Cancer ( PATTERN )
Status: Completed | Type: Observational
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Kerri Winters, Principal Investigator, OHSU Knight Cancer Institute
Other Study IDs: STUDY00021969; NCI-2021-05944 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00021969 (Other: OHSU Knight Cancer Institute); R01CA248059 (NIH)
Record Dates: First submitted 2023-02-23; First posted 2023-03-30 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Hematopoietic and Lymphoid Cell Neoplasm; Malignant Solid Neoplasm
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational (survey, assessment, SmartSocks, monitor): Patients complete surveys and clinic assessments at baseline, every 4-6 weeks during chemotherapy, and then every 3 months for 1 year after completion of chemotherapy. Clinic assessments include tests of neuropathy, upper and lower body strength, balance, and mobility. Patients complete weekly symptom surveys and wear instrumented socks and an activity monitor at regular intervals at home during chemotherapy treatment and for 1 year after completion of chemotherapy. Patients' medical records are also reviewed. After main study, patients may optionally complete surveys every 6 months for up to 5 years on study.
  Interventions: Procedure: Assessment of Therapy Complications; Other: Electronic Health Record Review; Other: Medical Device Usage and Evaluation; Other: Survey Administration

INTERVENTIONS:
Procedure: Assessment of Therapy Complications — Complete clinic assessments
Other: Electronic Health Record Review — Medical records are reviewed
Other: Medical Device Usage and Evaluation — Wear SmartSocks
Other: Medical Device Usage and Evaluation — Wear activity monitor
Other: Survey Administration — Complete survey

SUMMARY:
This study investigates the effects of treatment from chemotherapy for cancer on symptoms, function, and falls during treatment and through the recovery phase of cancer care. The goal is to identify simple tests that can help medical providers predict which and when patients show increased risk for falls and functional decline and informing rehabilitation providers about which mobility deficits to target.

DETAILED DESCRIPTION:
Aggressive treatments for cancer have improved survival, but often cause serious long-term adverse effects on daily life that last for many years. Chemotherapy-induced peripheral neuropathy (CIPN) is a persistent cancer treatment-related symptom that may negatively impact physical functioning, falls, and quality of life.

The persistence of CIPN symptoms and their relationship with life-threatening falls and disability point to a gap in oncology and follow-up care. A critical first step toward filling this gap is to characterize the natural trajectories of symptoms, functioning, and falls across the in-treatment and recovery phases of cancer care.

This study will prospectively enroll 200 adults with cancer that are scheduled to receive neurotoxic chemotherapy at the Portland campus of Oregon Health & Science University, 5 OHSU Knight Cancer Institute community hematology-oncology clinics, and OHSU research affiliate sites. Data collection occurs at patients' routine clinical appointments and at home via electronic surveys and passive monitoring devices. In the clinic, data collection occurs at 4-6 week intervals during treatment according to each patient's infusion schedule, and then approximately every 3 months for an additional year during routine follow-up care. Clinic-based assessments include tests of perceived sensation (tuning fork, monofilament, and biothesiometer), upper body strength (handgrip dynamometry), lower body strength (chair stand test), static balance (postural sway), and dynamic balance (Timed Up and Go test). Non-clinic-based data collection occurs weekly and assesses symptoms and falls via web-based surveys. At time points corresponding to clinic testing visits, participants are sent home with passive monitoring devices (instrumented socks and wrist-worn activity monitors) that measure physical activity and mobility.

PRIMARY OBJECTIVE:

I. To characterize trajectories of chemotherapy induced peripheral neuropathy (CIPN) symptoms and physical functioning (physical activity, mobility, self-report functioning and disability) and capture the variability in different patient trajectories across treatment and one year of recovery among persons receiving neurotoxic chemotherapy for cancer.

SECONDARY OBJECTIVE:

I. Determine whether or not patient characteristics alone can predict symptom and functioning trajectories or if adding clinical factors and simple tests of mobility significantly improves predictive capacity.

OUTLINE:

Patients complete surveys and clinic assessments at baseline, every 4-6 weeks during chemotherapy, and then every 3 months for 1 year after completion of chemotherapy. Clinic assessments include tests of neuropathy, upper and lower body strength, balance, and mobility. Patients complete weekly symptom surveys and wear instrumented socks and an activity monitor at regular intervals at home during chemotherapy treatment and for 1 year after completion of chemotherapy. Patients' medical records are also reviewed.

ELIGIBILITY:
Inclusion Criteria:

* Age 40-85 years old on date of enrollment.
* Diagnosed with stage I-III cancer, or stage IV cancer considered curable, other than cancers or metastases in the brain or spinal cord.
* Scheduled to receive any neurotoxic chemotherapy including taxane derivative, platinum complex, and/or vinca alkyloids

Exclusion Criteria:

* Previously received neurotoxic chemotherapy
* Cognitive difficulties that preclude answering the survey questions, participating in the performance tests, or giving informed consent
* A medical condition, movement or neurological disorder, or medication use that contraindicates participation in mobility testing and/or that confounds the ability to detect treatment-related changes in balance and mobility. Specific medical conditions include, but are not limited to, severe dystrophy, severe spasticity, epilepsy, seizures, Alzheimer's and dementia, while physical conditions include a severe balance disorder (i.e., later-stage Parkinson's, stroke), inability to ambulate (use of an assistive device permitted), inability to stand for 3 minutes, or severe hearing or vision problem

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with stage I-III cancer without neurologic involvement who are scheduled to receive neurotoxic chemotherapy at Oregon Health & Science University (OHSU) Knight Cancer Institute
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2020-10-22 (Actual); Primary Completion 2025-06-06 (Actual); Study Completion 2025-06-06 (Actual)

PRIMARY OUTCOMES:
Change in patient-reported neuropathy | Baseline up to 1 year after completion of chemotherapy (average of 16 months)
  Measured using the neuropathy subscale of the Functional Assessment of Cancer Therapy - Gynecologic Oncology Group Neurotoxicity (FACT-GOG-NTX-13) questionnaire, which assesses the presence, severity and impact of neuropathy symptoms in patients receiving neurotoxic chemotherapy. The scale ranges from 0-52, with lower scores indicating worse quality of life due to neuropathy.
Change in patient-reported neuropathy | Baseline up to 1 year after completion of chemotherapy (average of 16 months)
  Measured using the Patient-Reported Outcomes version of the Common Toxicity Criteria and Adverse Events version 1.0 (PRO-CTCAE™) reporting tool. Two items from the PRO-CTCAE™ ask if the patient experienced numbness or tingling in the hands or feet in the last 7 days using a 5-pt scale (0=none to 4=very severe) and how much the symptom interfered with their daily life using a 5-pt scale (0=not at all to 4=very much).
Change in perceived disability | Baseline up to 1 year after completion of chemotherapy (average of 16 months)
  Measured using the disability component of the Late-Life Function and Disability Instrument (LLFDI) which assesses disability in terms of frequency and limitation in performing 16 life tasks. Scores range from 0 to 100, with higher scores indicating less disability.
Change in daily functional mobility | Baseline up to 1 year after completion of chemotherapy (average of 16 months)
  Measured using instrumented socks (APDM.com) with inertial sensors embedded into neoprene ankle wraps. Patients wear the instrumented socks during waking hours over 7-day periods that correspond to each in-clinic assessment.
Change in daily physical activity | Baseline up to 1 year after completion of chemotherapy (average of 16 months)
  Measured using ActiGraph GT9X Link devices. The ActiGraph algorithms generate accurate and reliable data on total energy expenditure (kcal/d). Patients wear the devices over 7-day periods that correspond to each in-clinic assessment.

SECONDARY OUTCOMES:
Falls | Baseline up to 1 year after completion of chemotherapy (average of 16 months)
  Falls over the past 12 months will be assessed retrospectively at baseline and prospectively at weekly intervals using in-house surveys. These surveys ask subjects about the number of falls, the number of injurious falls, and medical care resulting from a fall during the observation period.
Change in quality of life | Baseline up to 1 year after completion of chemotherapy (average of 16 months)
  Measured using the European Organization for Research and Treatment of Cancer - Quality of Life Questionnaire for Cancer (EORTC-QLQ-C30). Global quality of life and subdomains of quality of life are scored from 0-100, with higher scores indicating better quality of life.
Change in patient-reported symptoms | Baseline up to 1 year after completion of chemotherapy (average of 16 months)
  Assessed weekly with the Patient Reported Outcomes - Common Terminology Criteria for Adverse Events (PRO-CTCAE™) reporting tool items. The PRO-CTCAE™ uses 5-pt scales to assess the severity (0=none to 4=very severe), frequency (0=never to 4=almost constantly), and interference (0=not at all to 4=very much) of symptoms in daily life within the previous 7 days.
Change in objective loss of perceived sensation | Baseline up to 1 year after completion of chemotherapy (average of 16 months)
  Measured using a tuning fork test.
Change in objective loss of perceived sensation | Baseline up to 1 year after completion of chemotherapy (average of 16 months)
  Measured using biothesiometry.
Change in upper extremity strength | Baseline up to 1 year after completion of chemotherapy (average of 16 months)
  Measured by handgrip dynamometry.
Change in static balance | Baseline up to 1 year after completion of chemotherapy (average of 16 months)
  Measured by a postural sway test that assesses how well a person maintains their balance during 30 seconds of quiet standing using Mobility Lab sensors and software (APDM.com). Increased sway indicates poor balance control and is associated with increased risk of falls.
Change in functional mobility | Baseline up to 1 year after completion of chemotherapy (average of 16 months)
  Measured by the Timed Up and Go (TUG) test. The TUG test evaluates the time that it takes a person to rise from a chair, walk 3 meters, then turn around and return to the chair in a seated position. Slower TUG times are associated with an increased risk of falls and disability.
Change in objective functional strength | Baseline up to 1 year after completion of chemotherapy (average of 16 months)
  Measured by a timed chair stand test (seconds required to rise from a chair 5 times). Chair stand time >12 seconds has been shown to predict a 2.4 increased risk of falls in older adults.
Change in skeletal muscle index | Baseline up to 1 year after completion of chemotherapy (average of 16 months)
  Clinically acquired abdominal and thoracic computed tomography images will be segmented into fat and lean tissue compartments according to their non-overlapping radiodensity ranges. Skeletal muscle index is calculated as skeletal muscle cross-sectional area divided by height in meters squared.

CONTACTS AND LOCATIONS:
Overall Officials: Kerri Winters-Stone, Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States

REFERENCES:
- [Derived] Winters-Stone KM, Krasnow SM, Horak FB, Mancini M, Cameron MH, Dieckmann NF, Stoyles SA, Roeland EJ. Identifying trajectories and predictors of chemotherapy-induced peripheral neuropathy symptoms, physical functioning, and falls across treatment and recovery in adults treated with neurotoxic chemotherapy: the PATTERN observational study protocol (NCT05790538). BMC Cancer. 2023 Nov 10;23(1):1087. doi: 10.1186/s12885-023-11546-2. PMID 37946117